CLINICAL TRIAL: NCT06197360
Title: Effects of a Health Education Intervention Based on the Behaviour Change Wheel on Fear of Hypoglycemia in Patients With Type 2 Diabetes Mellitus: a Pilot Study
Brief Title: Effects of a Health Intervention on Fear of Hypoglycemia : a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhao Yueqi, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YZUHL20210088
Record Dates: First submitted 2023-12-21; First posted 2024-01-09 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus; Fear of Hypoglycemia; Health Education; Impaired Awareness of Hypoglycemia; Self-Management
Keywords: Type 2 Diabetes Mellitus; Fear of hypoglycemia; Behavior Change Wheel theory; Impaired Awareness of Hypoglycemia; Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General diabetes health education (Placebo Comparator): Patients were provided with regular medication guidance, dietary guidance, exercise guidance and popularization of related diabetes knowledge; regular daily blood glucose testing and recording; and timely answers to patients' clinical problems and psychological support.
  Interventions: Behavioral: General diabetes health education
- Based on BCW Theory of Health Education (Experimental): A FOH intervention program based on BCW theory was implemented on top of the control group.
  Interventions: Behavioral: Based on BCW Theory of Health Education

INTERVENTIONS:
Behavioral: Based on BCW Theory of Health Education — Questionnaire collection, face-to-face interview, and interpretation of the manual on the first day of admission; diabetes self-management teaching on the second day; and hypoglycemia-related lectures and hands-on teaching on the fourth day. Day 6 hypoglycemia fear case discussion. Face-to-face teaching and formulation of blood glucose management plan on the first day before discharge; WeChat push or telephone return visit one week and two weeks after discharge; WeChat push, telephone return visit and questionnaire collection three weeks after discharge.
  Arms: Based on BCW Theory of Health Education
Behavioral: General diabetes health education — Patients were provided with regular medication guidance, dietary guidance, exercise guidance and popularization of related diabetes knowledge; regular daily blood glucose testing and recording; and timely answers to patients' clinical problems and psychological support.
  Arms: General diabetes health education

SUMMARY:
The purpose of this study was to construct a Fear of Hypoglycemia(FoH) intervention program for type 2 diabetic patients based on the Behaviour Change Wheel (BCW) theory and to investigate the feasibility, acceptability, and initial effects of the program.

DETAILED DESCRIPTION:
In this study, eligible participants were randomized in a 1:1 ratio into an intervention group (health education based on BCW theory given on top of regular diabetes health education) and a control group (regular diabetes health education), with a 4-week intervention period and a 4-week follow-up period, for a total of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the 2020 Chinese guidelines for the prevention and treatment of type 2 diabetes mellitus
* Age ≥18 years
* Duration of diabetes mellitus ≥1 year
* FOH according to the elevated item endorsement criterion (E I criterion): ≥3 points on any item of the Hypoglycemic Fear-Worry Scale (HFS-WS)
* Patients who have the ability to listen, read, write, walk, and cooperate to complete the study
* Patients who have a smart phone, and can skillfully use WeChat or telephone to communicate
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients with comorbid acute complications or other serious diseases or disorders of consciousness, such as diabetic hypertonic state, tumors, coma, etc.
* Patients with comorbid psychiatric diseases or taking psychotropic drugs
* Patients who have recently or are participating in other studies on similar topics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueqi Zhao, Bachelor, Principal Investigator — Yangzhou University
Locations (1):
- Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
No plans to provide IPD.

REFERENCES:
- [Result] Zhong W, Lin L, Gong X, Chen Z, Chen Y, Yan S, Zhou Y, Zhang X, Hu H, Tong L, Cheng C, Gu Q, Chen Y, Yu X, Huang Y, Yuan C, Lou M; MISSION investigators. Evaluation of a multicomponent intervention to shorten thrombolytic door-to-needle time in stroke patients in China (MISSION): A cluster-randomized controlled trial. PLoS Med. 2022 Jul 5;19(7):e1004034. doi: 10.1371/journal.pmed.1004034. eCollection 2022 Jul. PMID 35788767
- [Derived] Zhao Y, Zhang L, Pang J, Qiu J, He Y, Xu Z, Han M, Liu L, Wan X, Wang J, Zhang Y. Effects of a health education intervention based on the behavior change wheel on fear of hypoglycemia behavior in type 2 diabetes mellitus patients: a randomized controlled pilot trial. Acta Diabetol. 2025 Dec;62(12):2071-2084. doi: 10.1007/s00592-025-02549-5. Epub 2025 Jun 23. PMID 40548996

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Declined to participate (n= 11) Too busy (n= 3) Too sick (n= 2) Not interested (n= 6)
Period: Overall Study
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 7 | 11 | 18
  >=65 years | 16 | 13 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 9 | 10 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 25 | 25 | 50
BMI（kg/m^2) [Count of Participants; unit: Participants]
  <18.5 | 1 | 1 | 2
  18.5~23.9 | 14 | 19 | 33
  24~28 | 6 | 5 | 11
  ≥28 | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Fear Behavioral
Description: Hypoglycemia Fear Survey - Behavior Scale consists of 19 entries and is scored on a 5-point Likert scale from 1 to 5, with total scores ranging from 15 (lowest) to 95 (highest), with the higher scores indicating that the patients' hypoglycemia fear-behavior is more pronounced, and the higher the level of fear of hypoglycemia.
Time Frame: Baseline, immediately after the intervention and after the 4 weeks follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 59.60 (11.61) | 63.88 (11.63)
  Immediately after the intervention | 57.52 (12.33) | 44.20 (5.59)
  After the 4 weeks follow-up | 55.16 (10.68) | 39.72 (5.34)

2. Primary Outcome: Hypoglycemia Fear Worry
Description: Hypoglycemic fear Survey - Worry Scale was used to evaluate the patients' hypoglycemic feelings in the past 6 months. There were 13 items in the scale, using 5-point Likert scale, with scores ranging from low to high 0-4, and the total score ranging from 0 (lowest) to 52 (highest). The higher the score, the higher the patient's fear of hypoglycemia.
Time Frame: Baseline, immediately after the intervention and after the 4 weeks follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 32.72 (4.09) | 32.96 (2.89)
  Immediately after the intervention | 29.76 (2.64) | 18.76 (3.63)
  After the 4 weeks follow-up | 27.16 (4.15) | 15.44 (3.38)

3. Secondary Outcome: Gold Rating
Description: Gold Score was first proposed by Professor Gold in the UK in 1994. It is the most commonly used assessment method for Impaired Awareness of Hypoglycemia, which reflects patients' awareness of hypoglycemia at the same time. The only question with this approach is, "Do you know when your low blood sugar started?" Likert scores 7 on a scale of "1" (always aware) to "7" (never aware), with an overall score from 1 (lowest) to 7 (highest). An overall score of 1-3 is considered normal hypoglycemic self-awareness, and a score of ≥4 indicates the presence of IAH.
Time Frame: Baseline, immediately after the intervention and after the 4 weeks follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 2.84 (1.28) | 2.88 (1.26)
  Immediately after the intervention | 2.32 (1.07) | 1.68 (0.69)
  After the 4 weeks follow-up | 1.84 (0.90) | 1.28 (0.46)

4. Secondary Outcome: The Patients Assessment Chronic Illness Care( PACIC)
Description: The Patient Assessment Chronic Care Scale was developed with support from the Johnson Foundation to assess the quality of care provided by healthcare organizations. Patients use this scale to report their perceived level of medical support. The PACIC scale consists of five dimensions and 20 questions, each of which is rated on a 5-point Likert scale (1 to 5), with higher scores (close to 5) indicating greater support from healthcare professionals. The score for each dimension is calculated based on the average score of the items it contains, and the total table score is calculated based on the average score of all 20 items, with a minimum score of 1 and a maximum score of 5. Total scale score ≤1.75 is classified as low level of medical support; An overall average score of 1.75 to 3.5 indicates moderate medical support; Total mean score ≥3.5 was classified as high medical support.
Time Frame: Baseline, immediately after the intervention and after the 4 weeks follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.42 (0.45) | 3.40 (0.45)
  Immediately after the intervention | 3.69 (0.34) | 4.45 (0.26)
  After the 4 weeks follow-up | 3.55 (0.41) | 4.46 (0.21)

5. Secondary Outcome: The Self-management Attitude Scale for Diabetes Patients
Description: The Self-Management Attitude Scale for Diabetic Patients is a sub-scale of the Self-Management Knowledge, Attitude and Behavior Assessment Scale for Diabetic Patients compiled by the Chinese Center for Prevention and Control of Chronic Noncommunicable Diseases (CPCNCD). The scale included five items that assessed patients' attitudes toward diabetes health education, diet control, physical activity, medication adherence, and blood glucose monitoring. The 5-point Likert scale was used, with 1 indicating "very important" and 5 indicating "very unimportant", and the scores were divided into 0.2, 0.4, 0.6, 0.8 and 1.0 in order from low to high. The total score of the five items is the total self-management attitude score (range 1-5), and a score below 3.0 indicates a poor self-management attitude. A score of 3.0 to 4.25 indicates an average self-management attitude, while a score of 4.25 or above indicates a good self-management attitude.
Time Frame: Baseline, immediately after the intervention and after the 4 weeks follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.91 (0.68) | 4.10 (0.58)
  Immediately after the intervention | 4.21 (0.53) | 4.78 (0.18)
  After the 4 weeks follow-up | 4.28 (0.45) | 4.83 (0.19)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Evaluated through standardized questionnaires, regular assessments by researchers, and periodic laboratory inspections. No participants experienced adverse events.
Arm/Group | General Diabetes Health Education | Based on BCW Theory of Health Education
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT06197360/Prot_SAP_000.pdf